CLINICAL TRIAL: NCT03316859
Title: A Prospective Randomized, Double-Blind Study to Evaluate the Addition of Naloxegol to the Pre-Op Regimen of the Cardiac Surgery Patient and Its Effect on Opioid-Induced Constipation
Brief Title: Naloxegol and Opioid-induced Constipation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-020
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-06

CONDITIONS: Constipation; Constipation Drug Induced
Keywords: opioid-induced constipation (OIC)
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Naloxegol (Experimental): naloxegol 25 mg pill
  Interventions: Drug: Naloxegol 25 MG
- Placebo (Placebo Comparator): placebo pill
  Interventions: Other: Placebo pill

INTERVENTIONS:
Drug: Naloxegol 25 MG — Naloxegol 25 mg administered 1 hour pre-operatively
  Other Names: Movantik
  Arms: Naloxegol
Other: Placebo pill — Placebo pill administered 1 hour pre-operatively
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial to examine the effectiveness of adding one 25mg dose of naloxegol to the cardiac surgery pre-operative regimen.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled trial to examine the effectiveness of adding one 25mg dose of naloxegol to the cardiac surgery pre-op regimen. There will be 140 subjects per study group. The patient and treating physician/nurse will be blinded as to which group the subject is assigned. On the day of surgery, subjects in both groups will complete a questionnaire to assess compliance with prescribed pre-operative regimen. Subjects in both groups will receive post-operative bowel regimen in the cardiovascular intensive care unit (CVICU) according to current standard of care, including procedures for rescue medications for constipation prevention and induction of a bowel movement.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective cardiac surgery at Bethesda North TriHealth Hospital
* Admitted to Bethesda North TriHealth Hospital CVICU post-surgery

Exclusion Criteria:

* Medically unstable
* Cognitive deficits that impair the patient's ability to understand the informed consent
* Language barriers
* Patient has a documented diagnosis of one of the following: Crohn's disease; Ulcerative Colitis; History of bowel surgery that will impact absorption of study drug (as deemed by physician); History of small bowel obstruction
* Chronic constipation requiring subject to take one of the following medications on a daily basis prior to time of consent: Linzess, Trulance, Amitza, Senna/Senokot, Colace, Dulcolax, Miralax, Metamucil
* Patients on following medications prior to time of consent: Diltiazem, Verapamil, Amiodarone, Ketoconazole, Clarithromycin/ erythromycin, Antivirals
* Conditions that present an increased risk of bowel perforation (as determined by the physician)
* Pre-existing diagnosis of opioid-induced constipation AND receiving naloxegol as a treatment by their physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to substantial bowel movement | Post-operative day 1
  Time to bowel movement of Type 2 or higher on the Bristol stool chart
Time to substantial bowel movement | Post-operative day 2
  Time to bowel movement of Type 2 or higher on the Bristol stool chart
Time to substantial bowel movement | Post-operative day 3
  Time to bowel movement of Type 2 or higher on the Bristol stool chart
Time to substantial bowel movement | Post-operative day 4
  Time to bowel movement of Type 2 or higher on the Bristol stool chart
Time to substantial bowel movement | Post-operative day 5
  Time to bowel movement of Type 2 or higher on the Bristol stool chart

SECONDARY OUTCOMES:
Rescue medications | Post-operative day 1
  Amount of rescue medications
Rescue medications | Post-operative day 2
  Amount of rescue medications
Rescue medications | Post-operative day 3
  Amount of rescue medications
Rescue medications | Post-operative day 4
  Amount of rescue medications
Rescue medications | Post-operative day 5
  Amount of rescue medications

OTHER OUTCOMES:
Length of stay | Post-operative day 1
  CVICU length of stay
Length of stay | Post-operative day 2
  CVICU length of stay
Length of stay | Post-operative day 3
  CVICU length of stay
Length of stay | Post-operative day 4
  CVICU length of stay
Length of stay | Post-operative day 5
  CVICU length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Scott McCardle, MD, Principal Investigator — Bethesda North TriHealth Hospital
Locations (1):
- Bethesda North TriHealth Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chey WD, Webster L, Sostek M, Lappalainen J, Barker PN, Tack J. Naloxegol for opioid-induced constipation in patients with noncancer pain. N Engl J Med. 2014 Jun 19;370(25):2387-96. doi: 10.1056/NEJMoa1310246. Epub 2014 Jun 4. PMID 24896818
- [Background] DePriest AZ, Miller K. Oxycodone/Naloxone: role in chronic pain management, opioid-induced constipation, and abuse deterrence. Pain Ther. 2014 Jun;3(1):1-15. doi: 10.1007/s40122-014-0026-2. Epub 2014 May 6. PMID 25135384
- [Background] Nelson AD, Camilleri M. Chronic opioid induced constipation in patients with nonmalignant pain: challenges and opportunities. Therap Adv Gastroenterol. 2015 Jul;8(4):206-20. doi: 10.1177/1756283X15578608. PMID 26136838